CLINICAL TRIAL: NCT00030524
Title: A Phase II Clinical, Biological and Pharmacological Study of ZD1839 in Patients With Advanced Colorectal Carcinoma Refractory to 5-Fluorouracil (5-FU) and Irinotecan Chemotherapy
Brief Title: ZD 1839 in Treating Patients With Locally Advanced or Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000069174; UTHSC-0015011185; SACI-IDD-01-01; NCI-3753
Record Dates: First submitted 2002-02-14; First posted 2003-05-07 (Estimated); Last update posted 2012-10-30 (Estimated); Status verified 2012-10

CONDITIONS: Colorectal Cancer
Keywords: stage III colon cancer; stage IV colon cancer; stage III rectal cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer; adenocarcinoma of the colon; adenocarcinoma of the rectum
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Gefitinib

INTERVENTIONS:
Drug: gefitinib

SUMMARY:
RATIONALE: Biological therapies such as ZD 1839 may interfere with the growth of tumor cells and slow the growth of colorectal cancer.

PURPOSE: Phase II trial to study the effectiveness of ZD 1839 in treating patients who have locally advanced or metastatic colorectal cancer that has not responded to chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the progression-free rate at 16 weeks, response rate, time to treatment failure, and survival of patients treated with gefitinib for locally advanced or metastatic colorectal adenocarcinoma that is refractory to fluorouracil, irinotecan, and capecitabine.
* Correlate the pharmacodynamic effects of this drug with indices of clinical benefit (e.g., tumor growth inhibition, time to tumor progression, and survival) in these patients.
* Determine whether the status of epidermal growth factor receptor activation and signaling are predictive of clinical outcome in patients treated with this drug.

OUTLINE: This is a multicenter study.

Patients receive oral gefitinib once daily. Treatment continues every 28 days in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 18-46 patients will be accrued for this study within 5-12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed colorectal adenocarcinoma

  * Metastatic or locally advanced disease
  * Not amenable to curative therapy
* Documentation of disease progression within the past 6 months
* Previously treated with fluoropyrimidine- and irinotecan-based chemotherapy (including capecitabine) administered either concurrently (no more than 2 regimens) or sequentially (no more than 3 regimens) for advanced disease
* At least 1 unidimensionally measurable lesion

  * At least 20 mm by conventional techniques OR at least 10 mm by spiral CT scan
* No known brain metastases

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2 OR
* Karnofsky 60-100%

Life expectancy:

* More than 12 weeks

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* AST/ALT no greater than 3 times ULN (5 times ULN if liver metastasis present)

Renal:

* Creatinine no greater than 1.5 times ULN OR
* Creatinine clearance at least 60 mL/min

Cardiovascular:

* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia

Ophthalmic:

* No significant ophthalmic conditions, including:

  * Severe dry-eye syndrome
  * Keratoconjunctivitis sicca
  * Sjogren's syndrome
  * Severe-exposure keratopathy
  * Disorders that may increase the risk for epithelium-related complications (e.g., bullous keratopathy, aniridia, severe chemical burns, or neutrophilic keratitis)

Other:

* Able to take oral gefitinib
* No other uncontrolled concurrent illness
* No ongoing or active infection
* No psychiatric illness or social situation that would preclude study participation
* No prior gastrointestinal disorders (e.g., malabsorption syndrome)
* No prior allergic reactions attributed to compounds of similar chemical or biological composition to gefitinib
* No other prior malignancy except carcinoma in situ of the cervix, nonmelanoma skin cancer, or other cancer from which the patient has been free of evident disease for more than 5 years and/or has less than a 20-30% estimated likelihood of recurrence
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* See Disease Characteristics
* At least 30 days since prior chemotherapy and recovered

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* No prior gastric resection

Other:

* No other prior therapy for advanced disease
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No other concurrent investigational or commercial agents or therapies for the malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-01; Primary Completion 2003-09 (Actual); Study Completion 2003-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chris H. Takimoto, MD, PhD, Study Chair — The University of Texas Health Science Center at San Antonio
Locations (2):
- United States (2):
  - Institute for Drug Development, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas